CLINICAL TRIAL: NCT01365351
Title: Non-interventional Study With ZOMACTON in Children With Growth Hormone Deficiency
Brief Title: Online Surveillance of Treatment of Children With Growth Hormone Deficiency With ZOMACTON
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Ferring Arzneimittel GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: ZOM/011207/03
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Growth hormone: Children with growth hormone deficiency
  Interventions: Other: Growth hormone

INTERVENTIONS:
Other: Growth hormone — Drug given by prescription

SUMMARY:
The purpose of this study is to investigate long-term treatment with Zomacton® for pituitary short stature in children with insufficient growth hormone production and/or short stature caused by Turner syndrome.

ELIGIBILITY:
Inclusion Criteria:

* therapeutic need according to SPC
* written informed consent

Exclusion Criteria:

* contraindications according to SPC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinics and private practices
Sampling Method: Non-Probability Sample
Enrollment: 1034 (Actual)
Dates: Start 2007-12-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of ZOMACTON | Up to 5 years
  measured by: body height, increase of body height per annum

SECONDARY OUTCOMES:
Efficacy measured by further parameters | Up to 5 years
  measured by: weight, increase weight per annum sitting height, increase of sitting height per annum head circumference per annum bone age, increase of bone age per annum puberty development IGF-1, IGFBP-3 psychological cofactors
Safety of Zomacton and application device | Up to 5 years
  measured by: local adverse reactions to the application device adverse events of Zomacton safety laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (58):
- Germany (58):
  - Investigational Site, Konrad-Adenauer-Allee 33, Augsburg
  - Investigational Site, Friedrichstr. 36-42, Dresden
  - Investigational Site, Blücherstr. 4, Erfurt
  - Investigational Site, Loschgestr. 15, Erlangen
  - Investigational Site, Düsseldorfer Str. 1-7, Frankfurt (Main)
  - Investigational Site, Stresemannallee 1-3, Frankfurt (Main)
  - Investigational Site, Wilhelm-Breckow-Allee 20, Gummersbach
  - Investigational Site, Seminarstr. 2, Heidelberg
  - Investigational Site, Koblenzer Str. 115-155, Koblenz
  - Investigational Site, Elisenstr. 12, Oldenburg
  - Investigational Site, Elisabethenstr. 15, Ravensburg
  - Investigational Site, Chausseestr. 119, State of Berlin
  - Investigational Site, Marienstr. 6-8, Vechta
  - Investigational Site, Geranienweg 7, Bad Langensalza
  - Investigational Site, Augustenburger Platz 1, Berlin
  - Investigational Site, Chausseestraße 119, Berlin
  - Investigational Site. Gotlindestraße 2 - 20, Berlin
  - Investigational Site, Burgsteig 13, Bielefeld
  - Investigational Site, Alexandrinenstraße 5, Bochum
  - Investigational Site, Alter Markt 4, Bochum
  - Investigational Site, Flemmingstraße 4, Chemnitz
  - Investigational Site, Kerpener Str. 62 (Haus 26), Cologne
  - Investigational Site, Dr.-Friedrich-Steiner-Straße 5, Datteln
  - Investigational Site, Fetscherstraße 74, Dresden
  - Investigational Site, Hospitalstraße 44, Düren
  - Investigational Site, Düsseldorfer Straße 8, Düsseldorf
  - Investigational Site, Hufelandstraße 55, Essen
  - Investigational Site, Lyoner Straße 54, Frankfurt am Main
  - Investigational Site, Mathildenstraße 1, Freiburg im Breisgau
  - Investigational Site, Pippinplatz 4, Gauting
  - Investigational Site, Am Markt 3, Gehrden
  - Investigational Site, Robert-Koch-Straße 40, Göttingen
  - Investigational Site, Ernst-Grube-Straße 40, Halle
  - Investigational Site, Bleickenallee 38-40, Hamburg
  - Investigational Site, Lornsenstraße 4-6, Hamburg
  - Investigational Site, Werlerstraße 130, Hamm
  - Investigational Site, Brabeckstraße 153, Hanover
  - Investigational Site, Im Neuenheimer Feld 430, Heidelberg
  - Investigational Site, Seminarstraße 2, Heidelberg
  - Investigational Site, Kirrberger Straße, Homburg
  - Investigational Site, Kochstraße 2, Jena
  - Investigational Site, Ettlinger Straße 27, Karlsruhe
  - Investigational Site, Schwanenweg 20, Kiel
  - Investigational Site, Lutherplatz 40, Krefeld
  - Investigational Site, Johannisplatz 1, Leipzig
  - Investigational Site, Liebigstraße 20 a, Leipzig
  - Investigational Site, Birkenallee 34, Magdeburg
  - Investigational Site, Leipziger Straße 44, Magdeburg
  - Investigational Site, Kölner Platz 1, München
  - Investigational Site, Lindwurmstraße 4, München
  - Investigational Site, Promenadeplatz 12, München
  - Investigational Site, Albert-Schweitzer-Straße 33, Münster
  - Investigational Site, Helmut-Just-Straße 6, Neubrandenburg
  - Investigational Site, St.-Johannis-Mühlgasse 19, Nuremberg
  - Investigational Site, Dr.-Eden-Straße 10, Oldenburg
  - Investigational Site, Hauptkanal rechts 75, Papenburg
  - Investigational Site, Pettenkoferstraße 10, Rosenheim
  - Investigational Site, Eythstraße 24, Ulm